CLINICAL TRIAL: NCT06848829
Title: Difference of Tear Ferning Between Pre-and Post-menopausal Women and Between Post-menopausal Women with or Without Hormone Replacement Therapy (HRT)
Brief Title: Difference of Tear Ferning Between Women with and Without Menopausal.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chung Shan Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202400071B0
Record Dates: First submitted 2025-02-14; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye diagnosis; Tear ferning; menopause
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pre-manepausal women (No Intervention): Collect clinical information, tear and blood samples from women pre-menopause with dry eye syndrome.
- Post-manepausal women (Other): Collect clinical information, tear and blood samples from women post-menopause with dry eye syndrome.
  Interventions: Other: Pre-manepausal women

INTERVENTIONS:
Other: Pre-manepausal women — Compare tear ferning structure between pre-menopause and post-menopause women.
  Other Names: Post-manepausal women
  Arms: Post-manepausal women

SUMMARY:
Application of tear ferning test for clinical dry eye diagnosis and menopause

DETAILED DESCRIPTION:
Analyzing the difference in tear ferning structure between women pre and post-menopause with and without hormone replacement therapy (HRT). Tear and blood samples were collected for a menopause-related Enzyme-linked immunosorbent assay. Tear volume, tear osmolarity, intraocular pressure, and tear break-up time were also measured for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 65 years

Exclusion Criteria:

* No evident ocular diseases such as cornea, cataracts, vitreous degeneration, glaucoma, and retinopathy.
* Belong to vulnerable groups(pregnancy woman, prisoner, ethical minorities, economic or educationally disadvantaged subjects, disabled individuals such as those at terminal stage of tumorigenesis, blindness, terminal ill individuals)

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Schirmer's test | 5 minutes
  To assess tear secretion volume
Tear film breakup time | 20 seconds
  To assess tear quality
Ocular surface status | 3 minutes
  To assess ocular surface health status with lissamine green stain, health or corneal abrasion.
Tear ferning | 30 minutes
  crystal structure formed from tear drops on a slide be scored.
Menopause related hormone Enzyme-linked immunosorbent assay (ELISA) | 3 hours
  To assess FSH/LH/E2/Progesterone/Mc5AC/Lactoferrin concentration between pre- and post-manopause women.

SECONDARY OUTCOMES:
Ocular surface disease index | 20 minutes
  A questionnaire to assess the health status on ocular surface
  A final score is calculated which ranges from 0 to 100 with scores 0 to 12 representing normal, 13 to 22 representing mild dry eye disease, 23 to 32 representing moderate dry eye disease, and greater than 33 representing severe dry eye disease.
Intraocular pressure | 2 minutes
  To determine the effects of intervention on intraocular pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Jen-Ai Hospital, Taichung, Taiwan, Taiwan